CLINICAL TRIAL: NCT02475512
Title: A Total Body Wash Wipe Combined With a Genital Wipe Versus Standard Care (Water and pH Neutral Soap) for Washing of Incontinent Residents in a Long- Term Care Setting: a Multicenter Prospective Randomised Controlled Clinical Trial and Health Economical Analysis in Nursing Homes
Brief Title: Comparison of Wash Wipes and Standard Care in the Prevention of Incontinence-associated Dermatitis in Elderly
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, UCVV, University Centre for Nursing and midwifery, University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/0277; B670201524231 (Other: Ethics Committee UZ Gent)
Record Dates: First submitted 2015-05-21; First posted 2015-06-18 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Irritant Contact Dermatitis Due to Incontinence; Diaper Rash; Pressure Ulcer; Incontinence-associated Dermatitis
Keywords: elderly; long-term care
MeSH Terms: conditions — Diaper Rash; Pressure Ulcer | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wash wipes (Experimental): Washing with water and soap (standard care) will be replaced with two wash wipes during 30 days: (1) daily total body wash (using 3M Cavilon Bathing and Cleansing wipes) and (2) Continence Care (using 3M Cavilon Continence Care Wipes). No other preventive barrier or hydration products will be allowed in the genital-anal region.
  Interventions: Other: Wash wipes (3M)
- Standard care (Placebo Comparator): Washing will be done using water and pH neutral soap. No other preventive barrier or hydration products will be allowed in the genital-anal region.
  Interventions: Other: water and pH neutral soap

INTERVENTIONS:
Other: Wash wipes (3M)
  Other Names: 3M Cavilon Bathing & Cleansing Wipes; 3M Cavilon Continence Care Wipes
  Arms: Wash wipes
Other: water and pH neutral soap
  Arms: Standard care

SUMMARY:
Incontinence is a widespread problem in all health care setting. One of the main complications of incontinence is inflammation of the skin in the genital and anal region, also known as incontinence-associated dermatitis (IAD). IAD is a known risk factor of pressure ulcer development. Prevalence figures of IAD vary between 5.6% and 50%.

The primary aim of this study is to compare the effectiveness of a 3-in-1 genital wipe versus standard care (traditional water and soap) for the prevention of IAD. The second aim is to perform a health economic evaluation of the 3-in-1 genital wipe versus standard care, and third to compare the cost of a 2-in-1 total body wash wipe versus standard care for total body wash. Other outcomes are the comfort and tolerance of both the nurses and participants.

In this Randomized Controlled Trial, performed in 13 long-term care settings, the participants will undergo a 30 day study period. In the experimental intervention, the participants will be washed with body wash wipes and genital wipes. In the control group, the subjects will receive traditional care. IAD as well as Pressure Ulcer prevalence will be monitored. Subjective and objective time measurements will be performed.

ELIGIBILITY:
Inclusion Criteria:

* urinary incontinence, fecal incontinence or double incontinence
* depending on help for washing
* free of skin damage (without signs of pressure ulcers or IAD such as skin breakdown or redness)

Exclusion Criteria:

* not incontinent or minor incontinent (e.g. stress incontinence)
* urinary or fecal catheter
* use of incontinence wipes in the uro-genital area two weeks prior to the start of the study
* the use of a skin barrier product in the uro-genital area two weeks prior to screening
* presence of a bacterial/fungal infection in the uro-genital area

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 385 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence and category of Incontinence-Associated Dermatitis | within the first 30 days after start of the study

SECONDARY OUTCOMES:
Incidence and category of Pressure Ulcers | within the first 30 days after start of the study
Comfort and tolerance of the participant | On baseline, at day 14 and at day 30 (the end of the study)
  Questions on comfort and tolerance of the washing method will be assessed by the caregiver. At baseline (day 0) these questions will assess the traditional care. In the middle (day 14) and at the end of the study (day 30) the comfort and tolerance of washing with wash wipes will be assessed in the experimental group. In the control group, comfort and tolerance of traditional care will be assessed three times.
Comfort and preferences of the caregiver | On baseline, at day 14 and at day 30 (the end of the study)
  Questions on comfort and preferences of the washing method will be assessed. At baseline (day 0) these questions will assess the traditional care. In the middle (day 14) and at the end of the study (day 30) the comfort and preferences of washing with wash wipes will be assessed.
adverse effects of the intervention | within the first 30 days after start of the study
  Adverse effects such as skin irritation, rash, itching, treatment related pain, skin dryness related to the interventions under study will be monitored.
Cost of the experiment (use of wash wipes) versus the standard care | For the duration of the study (30 days)
  * recording the daily consumption of towels, wash wipes,...
  * subjective time analyses of the washing methods: Estimated time registration by the caregiver
  * objective time analyses of the washing methods: time registration using a chronometer, conducted by researcher
  * retrieval of overhead costs related to traditional hygienic care: washing equipment purchase costs, general water and electricity: given per institution

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, PhD, Principal Investigator — University Ghent
Locations (11):
- Belgium (11):
  - Woonzorgcentrum Sint-Jozef, Bruges
  - Woonzorgcentrum Ceder aan de Leie, Harelbeke
  - Woonzorgcentrum Heilig Hart, Kortrijk
  - Woonzorgcentrum Sint-Jozef, Kortrijk
  - Woonzorgcentrum De Samaritaan, Nukerke
  - Woonzorgcentrum de Boarebreker, Ostend
  - Woonzorgcentrum De Kroon, Sint-Gillis-Waas
  - Woonzorgcentrum Deken Darras, Tielt
  - Woonzorgcentrum Onze Lieve Vrouw van Lourdes, Wakken
  - Woonzorgcentrum Duneroze, Wenduine
  - Woonzorgcentrum Sint-Camillus, Wevelgem

REFERENCES:
- [Background] Beeckman D, Van Lancker A, Van Hecke A, Verhaeghe S. A systematic review and meta-analysis of incontinence-associated dermatitis, incontinence, and moisture as risk factors for pressure ulcer development. Res Nurs Health. 2014 Jun;37(3):204-18. doi: 10.1002/nur.21593. Epub 2014 Apr 3. PMID 24700170
- See also: Website of the research group — http://www.ucvvgent.be